CLINICAL TRIAL: NCT06795321
Title: Patients' Anesthesia Preferences for Cesarean Delivery: Exploring the Role of Personality Beliefs in Spinal vs. General Anesthesia
Brief Title: Personality and Anesthesia Preferences in Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Esra Turunc, Director, Ondokuz Mayıs University
Other Study IDs: PAPCD
Record Dates: First submitted 2025-01-18; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Cesarean Delivery; Personality Beliefs
Keywords: Cesarean delivery; Spielberger State Anxiety Inventory (STAI II); Personality Belief Questionnaire Short Form (PBQ-SF)
MeSH Terms: interventions — Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group S: spinal anesthesia
  Interventions: Procedure: Spinal anesthesia
- Group G: general anesthesia
  Interventions: Procedure: General anesthesia

INTERVENTIONS:
Procedure: Spinal anesthesia — Patients who preferred spinal anesthesia were included in this group.
  Groups: Group S
Procedure: General anesthesia — Patients who preferred spinal anesthesia were included in this group
  Groups: Group G

SUMMARY:
Cesarean deliveries (CD) under general anesthesia are still common despite higher risks. Clinical guidelines recommend neuraxial anesthesia, but many patients refuse it due to fear and anxiety. This study aims to compare the personality traits of mothers who chose general versus spinal anesthesia for CD.

DETAILED DESCRIPTION:
Cesarean deliveries (CD) under general anesthesia continue to be common in many countries, though the practice varies in frequency. In the United States, about 5.8% of CDs are performed under general anesthesia. In Europe, the rate is higher in some countries, with 10% in Germany, 30% in Spain, and 34% in the Czech Republic. The exact rate in the study's country is not known but is assumed to be high. Clinical guidelines suggest that neuraxial anesthesia (spinal or epidural) should be the preferred choice for CD unless there are specific contraindications. This recommendation stems from the increased risks of general anesthesia, which include airway complications, aspiration risks, significant blood loss, and the potential for intraoperative awareness.

General anesthesia may still be a suitable option when spinal anesthesia is contraindicated or in cases with severe complications such as fetal bradycardia, uterine rupture, heavy bleeding, or placental abruption. Despite these risks, many patients still choose or are administered general anesthesia, often rejecting neuraxial anesthesia. The use of general anesthesia for CD carries higher risks of anesthesia-related complications, surgical site infections, and venous thromboembolism. This highlights the need to minimize the unnecessary use of general anesthesia by better understanding the factors that influence patients' anesthesia preferences.

One of the most common reasons patients refuse regional anesthesia (spinal or epidural) is the fear of spinal injury, concerns about the pain from the needle insertion, or anxiety about witnessing the surgical procedure. On the other hand, those who opt for regional anesthesia often cite the fear of not waking up from general anesthesia and the desire to remain conscious during childbirth. Research also suggests that anxiety levels are linked to the choice of anesthesia, though previous studies have yielded conflicting results.

Study Hypothesis and Aim: The study hypothesizes that patients' anesthesia preferences during CD might be influenced by their personality traits. While no prior studies have examined the relationship between personality traits and anesthesia preferences specifically in CD patients, some studies have explored the impact of personality on maternal delivery preferences (whether a woman chooses CD or vaginal delivery). The primary aim of this study is to compare the personality belief scores of expecting mothers who undergo CD with either general or spinal anesthesia, according to their preferred anesthesia type.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 45 years,
* American Society of Anesthesiologists (ASA) classification of II-III,
* Who were planned to undergo elective cesarean delivery (CD)

Exclusion Criteria:

* Patients who did not agree to participate in the study
* Patients requiring emergency cesarean delivery (CD)
* Patients with an absolute contraindication to general or regional anesthesia
* Patients lacking the educational or mental capacity to complete the evaluation scales
* Patients who were not informed about the study during the preoperative visit or did not provide written consent to participate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Who were planned to undergo elective cesarean delivery (CD) (only female)
Study Population: Patients aged 18-45 years, classified as ASA II or III, admitted to the Gynecology and Obstetrics Clinic of Ondokuz Mayıs University Hospital and planned for elective cesarean delivery (CD) were included. The anesthesia method (general or spinal) was chosen at the patient's discretion.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Personality belief scores of patients who preferred general or spinal anesthesia | The time when the patients were in the preoperative waiting room before surgery.
  The personality belief was assessed using The Personality Belief Questionnaire Short Form (PBQ-SF). The Personality Belief Questionnaire Short Form (PBQ-SF) is a 65-item self-reported questionnaire designed to assess an individual's personality. The PBQ-SF was created by selecting the seven highest-scoring items for each personality trait from the original PBQ.12 The form contained statements related to ten different personality disorders/features (avoidant, dependent, passive-aggressive, obsessive-compulsive, antisocial, narcissistic, histrionic, schizoid, paranoid, and borderline). The patients were asked to rate the extent to which they agreed with these statements on a 0-4 scale (0 = not at all, 1 = slightly agree, 2 = moderately agree, 3 = very much agree, and 4 = totally agree). Personality traits were examined based on the scores generated by the responses. The PBQ-SF has been translated into Turkish and its validity.

SECONDARY OUTCOMES:
Patient satisfaction | postoperative day 1
  The patient were asked to evaluate their satisfaction with their anesthesia experience using a 4-point Likert scale (1 = poor, 2 = average, 3 = good, and 4 = very good).
Sociodemographic datas | preoperative 30 minutes ago
  patients' name, surname, age, education level, employment status, income level, previous pregnancy and anesthesia experiences, smoking habits, history of psychiatric illness, medication use, and factors influencing their anesthesia preference.
Spielberger State Anxiety Inventory (STAI I-II) | The time when the patients were in the preoperative waiting room before surgery.
  STAI is a 40-item self-report questionnaire that measures both state anxiety (how a person feels at the moment) and trait anxiety (how a person generally feels). It consists of two 20-item subscales, each scored on a 4-point scale, with scores ranging from 20 to 80. State anxiety is measured from "not at all" to "very much so," and trait anxiety from "almost never" to "almost always." The Turkish version was adapted in 1985, with higher scores indicating greater anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)

REFERENCES:
- [Derived] Turunc E, Bilgin S, Akdeniz S, Komurcu O, Tomak L, Ustun YB, Koksal E, Dost B. Patients' anesthesia preferences for Cesarean delivery: exploring the role of personality beliefs in spinal vs. General anesthesia. BMC Anesthesiol. 2025 Jul 1;25(1):313. doi: 10.1186/s12871-025-03185-w. PMID 40597644